CLINICAL TRIAL: NCT06234228
Title: Examining Bluetooth Haptic Device Use for Pain and Anxiety Reduction in Vascular Access Procedures
Acronym: VA+BHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 73750
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pain; Anxiety
Keywords: Vascular access
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BHD synced with mobile game (Experimental): At the beginning of the vascular access procedure, the BHD will be applied 5 cm above the needle insertion site and maintained in place throughout the procedure. It delivers a constant low-frequency vibration as well as tactile feedback from the game (GF).
  Interventions: Behavioral: BHD synced with mobile game
- BHD only (Other): The participant will wear the BHD 5 cm above the needle insertion site for the duration of the procedure. The BHD will deliver constant low-frequency vibration (CF).
  Interventions: Behavioral: Bluetooth Haptic Device (BHD)
- Standard of Care (No Intervention): The participant will not receive the BHD device. Participant will receive standard of care treatment.

INTERVENTIONS:
Behavioral: Bluetooth Haptic Device (BHD) — The BHD will deliver constant low-frequency vibration (CF).
  Arms: BHD only
Behavioral: BHD synced with mobile game — The BHD delivers a constant low-frequency vibration as well as tactile feedback from the game (GF).
  Arms: BHD synced with mobile game

SUMMARY:
This pragmatic, randomized study seeks to evaluate the applications of a novel vibrating device for reducing pediatric anxiety and distress during vascular access procedures.

ELIGIBILITY:
Inclusion Criteria:

* Between age 4-99
* Will undergo a vascular access procedure
* English speaking participant and parent or LAR

Exclusion Criteria:

* Legal guardian not present to obtain consent
* Child is unable to self-report pain or anxiety
* Child with a significant neurological condition, or major developmental disability
* Child with active infection of the hand or arm
* Major surgery within the last 48 hours

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2026-11-04 (Estimated)

PRIMARY OUTCOMES:
External observation for pain and anxiety using OBSD-r scale | during vascular access procedure
  OBSD-r contains 8-item scale assessing participant's affective state; Information Seeking, Crying, Screaming, Restraint, Verbal Resistance, Emotional Support, Verbal Pain and Flail.

SECONDARY OUTCOMES:
Faces Pain Scale-Revised for patients aged 4-11 | during vascular access procedure
  Detailed qualitative review of cognitive interview probes with question-by-question analysis of transcribed cognitive interviews to assess for basic comprehension and appropriate use of the FPS-R. This scale is measured from 0-10, where 0 = no pain and 10 = very much pain.
Numerical Rating Pain Scale (NRPS) for patients aged 12-17 | during vascular access procedure
  NRPS is a 11-point (0-10) Numeric Rating Pain Scale (NRPS), where 0 = no pain and 10 = worst possible pain.
modified induction compliance checklist (mICC) | during vascular access procedure
  The mICC score will be recorded by the trained research observers during the vascular access procedure. Perfect compliance (score of 0) was compared to those that lacked cooperation. mICC will be rated at the time of intervention and only requires one RA.
External observation for pain and anxiety using HRAD scale | during vascular access procedure
  HRAD contains 5-item scale assessing participant's affective state; happy, relaxed, anxious, distressed, with a yes/no answer to cooperation.
Children's Anxiety Meter-State (CAM-S) assessment | immediately before, immediately after vascular access procedure
  The CAM-S is completed by showing the child a picture of a mercury thermometer. This scale is measured from 1-10. Higher values indicate higher anxiety.
Self formulated procedural satisfaction survey (Patient and Parent) | immediately after vascular access procedure
  The survey contains 10 items and utilizes a 5-point Likert agreement scale with a score of 1 meaning "completely disagree" and 5 meaning "completely agree."
Self formulated procedural satisfaction survey (Healthcare provider) | immediately after vascular access procedure
  The survey contains 5 items and utilizes a 5-point Likert agreement scale with a score of 1 meaning "completely disagree" and 5 meaning "completely agree."

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Caruso, MD,PhD, Study Director — Stanford University
Locations (1):
- Lucile Packard Childrens Hospital Stanford, Palo Alto, California, United States